CLINICAL TRIAL: NCT06994455
Title: Efficacy of Local Doxycycline Gel Delivery Versus Doxycycline Nanoparticles Prepared Gel in The Treatment of Stage II Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: A020120230M
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1: doxycycline gel+SRP (Experimental): doxycycline gel (regular non-nanoparticle form) as an adjunct to mechanical debridement.
  Interventions: Procedure: scaling and root planing along with antibiotic intervention
- group 2: doxycycline-loaded(PLGA) nanoparticles gel +SRP (Experimental): doxycycline-loaded Poly lactic-co-glycolic acid (PLGA) nanoparticles gel as an adjunct to mechanical debridement.
  Interventions: Procedure: scaling and root planing along with antibiotic intervention
- group 3: mechanical debridement only. (Active Comparator): scaling and root planing alone
  Interventions: Procedure: scaling and root planing

INTERVENTIONS:
Procedure: scaling and root planing along with antibiotic intervention — doxycycline gel exhibits bacteriostatic activity against prevalent periodontal pathogens
  Arms: group 1: doxycycline gel+SRP
Procedure: scaling and root planing along with antibiotic intervention — the formulation of doxycycline and incorprating it with PLGA nano-particles will increase the absorption rate in gingival sulcus
  Arms: group 2: doxycycline-loaded(PLGA) nanoparticles gel +SRP
Procedure: scaling and root planing — control group in the study
  Arms: group 3: mechanical debridement only.

SUMMARY:
To evaluate the Efficacy of Local Doxycycline Gel Delivery Versus Doxycycline Nanoparticles Prepared Gel in The Treatment of stage II Periodontitis

Materials and methods: forty five patients (n=45) were selected from the Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mansoura University. 45 particpants are classified into 3 groups

Group 1(test group): 15 Patients will be treated with doxycycline gel (regular non-nanoparticle form) as an adjunct to mechanical debridement.

Group 2 (test group): 15 Patients will be treated with doxycycline-loaded Poly lactic-co-glycolic acid (PLGA) nanoparticles gel as an adjunct to mechanical debridement.

Group 3 (control group): 15 patients will be treated with mechanical debridement only.

After proper examination and diagnosis, full mouth supra- and subgingival scaling and root planning will be performed over two weeks (two consecutive days per week) and all periodontitis patients will be treated with ultrasonic scaler and hand instrument for meticulous removal of subgingival and supragingival plaque and calculus. All patients will receive oral hygiene instructions.

Gel Application:

After completion of scaling and root planning the doxycycline gel will be injected subgingivally in the deepest selected periodontitis pockets of the group 1 and doxycycline-loaded Poly lactic-co-glycolic acid (PLGA) gel in group 2 using a disposable syringe.

Care will be taken to apply the gel without traumatizing or damaging the periodontal tissues. Participants will be instructed to refrain from chewing hard or consuming sticky foods, brushing near the treated areas, or using any interdental aids for 1 week. The injection will be applied in the third week with maintenance of good oral hygiene.

Periodontal Parameters:

Changes in the clinical parameters will be evaluated. For all periodontitis patients, the Clinical assessment will be performed at baseline, after 4 weeks and after 8 weeks from the start of the study.

All these clinical parameters will be assessed:

1. Plaque Index according to Silness & Loe 1964.26
2. Gingival Bleeding Index according to Ainamo & Bay 1975.27
3. Probing pocket depth (PPD) 28 is measured from free gingival margin to the base of the pocket.
4. Clinical attachment level (CAL) 29 is measured from the cement-enamel junction to the base of the pocket.

Microbiological assessment:

Subgingival plaque sample collection will be done for semi-quantitative measuring of P.gingivalis and P.intermedia. Each periodontal site included in the study will be isolated with cotton rolls and dried with an air syringe to avoid contamination with saliva. Before sample collection, all clinically detected supragingival plaque are remove with a sterile curette to avoid contamination between supragingival and subgingival plaque. The subgingival plaque samples are collected by insertion of sterile medium size paper point into the pocket for 30 seconds. Samples with any saliva or blood contamination are discard. After that, the paper point is immediately store in a sterile microcentrifuge tube containing 1 ml of thioglycolate broth transport media and send immediately to microbial diagnostic and infection control unit (MDICU) for sample processing. Samples are culture anaerobically for detection of total bacterial count as well as p.gingivalis and p.intermedia count.

DETAILED DESCRIPTION:
Inclusion criteria: The selected patients included:

Patients of both sexes above 20 years old Patients with probing pocket depth ≤ 5 mm. No history of antibiotic and periodontal therapy in the last 3 months.

Exclusion criteria included:

Patients with systemic diseases. Pregnant and lactating females. Heavy smokers.

Gel Application:

After completion of scaling and root planning the doxycycline gel will be injected subgingivally in the deepest selected periodontitis pockets of the group

1, and doxycycline-loaded Poly lactic-co-glycolic acid (PLGA) gel in group 2 using a disposable syringe. Care will be taken to apply the gel without traumatizing or damaging the periodontal tissues. Participants will be instructed to refrain from chewing hard or consuming sticky foods, brushing near the treated areas, or using any interdental aids for 1 week. The injection will be applied in the third week with maintenance of good oral hygiene.

Microbiological assessment:

Subgingival plaque sample collection will be done for semi-quantitative measuring of P.gingivalis and P.intermedia. Each periodontal site included in the study will be isolated with cotton rolls and dried with an air syringe to avoid contamination with saliva. Before sample collection, all clinically detected supragingival plaque are remove with a sterile curette to avoid contamination between supragingival and subgingival plaque. The subgingival plaque samples are collected by insertion of sterile medium size paper point into the pocket for 30 seconds. Samples with any saliva or blood contamination are discard. After that, the paper point is immediately store in a sterile microcentrifuge tube containing 1 ml of thioglycolate broth transport media and send immediately to microbial diagnostic and infection control unit (MDICU) for sample processing. Samples are culture anaerobically for detection of total bacterial count as well as p.gingivalis and p.intermedia count.

Periodontal Parameters:

Changes in the clinical parameters will be evaluated. For all periodontitis patients, the Clinical assessment will be performed at baseline, after 4 weeks and after 8 weeks from the start of the study.

All these clinical parameters will be assessed:

1. Plaque Index according to Silness & Loe 1964.26
2. Gingival Bleeding Index according to Ainamo & Bay 1975.27
3. Probing pocket depth (PPD) 28 is measured from free gingival margin to the base of the pocket.
4. Clinical attachment level (CAL) 29 is measured from the cement-enamel junction to the base of the pocket.

Statistical Assessment:

Data will be analyzed using SPSS (statistical package for social sciences) version 28. Qualitative data will be presented as number and percent, Quantitative data will be tested for normality by Shapiro-Wilk test then described as mean and standard deviation for normally distributed data and median and range for non normally distributed. The appropriate statistical test will be applied according to data type with the following suggested tests: One Way ANOVA test and Kruskal Wallis test.

Patients eligible for this study will be screened by a comprehensive periodontal examination, and full periodontal charts will be obtained. Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017 AAP World Workshop

The patients will be informed about the treatment that they will receive and steps that will be done. This includes the possible effects or risks, and other treatment options according to the rules of the ethical committee of the Faculty of Dentistry, Mansoura University. The subjects must understand this explanation in broad terms. The subjects must be legally competent to give written consent before performing any required steps, proper case history. The research protocol will be presented on the ethical committee at faculty dentistry Mansoura university to get its approval.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes above 20 years old
* Patients with probing pocket depth ≤ 5 mm.
* No history of antibiotic and periodontal therapy in the last 3 months

Exclusion Criteria:

* Patients with systemic diseases.
* Pregnant and lactating females.
* Heavy smokers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-06-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
probing pocket depth reduction | 8 weeks
  pocket depth is calculated using periodontal probe to calculate the distance between the base of the pocket to the free gingival margin

SECONDARY OUTCOMES:
plaque index | 8 weeks
  according to Silness & Loe 1964
clinical attachment gain | 8 weeks
  measured from cemento-enamel junction to the base of the pocket
gingival bleeding index | 8 weeks
  according to Ainamo & Bay 1975
microbiological detection of p.gingivalis | 8 weeks
  Samples are culture anaerobically for detection p.gingivalis
microbiological detection for p.intermedia | 8 weeks
  Samples are culture anaerobically for detection p.intermedia

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura, Egypt, 35516, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided